CLINICAL TRIAL: NCT01501006
Title: Social and Behavioral Influences on Clinical Care
Brief Title: Social and Behavioral Influence (SBI)
Acronym: SBI
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ronald Epstein, Principal Investigator, University of Rochester
Other Study IDs: 33086; R01CA155376-01 (NIH)
Record Dates: First submitted 2011-11-30; First posted 2011-12-29 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Communication
Keywords: Physicians
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patient Roles: Physician communication styles will be evaluated with different patient roles.

SUMMARY:
The purpose of the study is to improve patient-physician communication and clinical decisions in the context of serious illness that may affect important clinical outcomes. The investigators will examine how variations in communication patterns and clinical decisions are affected by patient demographics (e.g age, sex), patient interactional style (e.g. communication behaviors) and physician characteristics (e.g. attitudes, background, training).

DETAILED DESCRIPTION:
This will be a randomized field experiment. Physicians will receive two unannounced covert standardized patient (SP) visits during the 12-24 months after enrollment. SPs are trained actors who will pose as patients to assess physician behavior and communication. Each SP will present just like a real patient, and will have a standardized fabricated scenario and identity. The SP visit will be unannounced; the physician will not be informed at the time of the visit that they are seeing an SP. The visits will be covertly audio-recorded. This is being conducted at 3 sites: University of Rochester, Rochester, NY; Purdue, IN; and University of Michigan.

ELIGIBILITY:
Inclusion Criteria:

* Currently in clinical practice
* Do not plan on moving during the next year

Exclusion Criteria:

* Non-physicians

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and Female physicians of all races and ethnicities
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2010-10; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Physicians Communication Style | 2 years
  To examine the degree to which physicians communication style (ex inclusive, authoritative) and clinical decisions (ex. aggressive,passive) differ according to patient characteristics. Unit of Measure: Audio recordings of office visits, will be transcribed, deidentified, and coded.

SECONDARY OUTCOMES:
Physician Communication Moderators (Sex,Class) | 2 years
  To examine how patients participating in their care reduces these patient-specific differences in physician communication behaviors and decisions. Unit of Measure: Audio recordings of office visits, will be transcribed, deidentified, and coded.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Epstein, MD, Principal Investigator — University of Rochester
Locations (1):
- University Of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Shields CG, Griggs JJ, Fiscella K, Elias CM, Christ SL, Colbert J, Henry SG, Hoh BG, Hunte HER, Marshall M, Mohile SG, Plumb S, Tejani MA, Venuti A, Epstein RM. The Influence of Patient Race and Activation on Pain Management in Advanced Lung Cancer: a Randomized Field Experiment. J Gen Intern Med. 2019 Mar;34(3):435-442. doi: 10.1007/s11606-018-4785-z. Epub 2019 Jan 10. PMID 30632104
- [Derived] Elias CM, Shields CG, Griggs JJ, Fiscella K, Christ SL, Colbert J, Henry SG, Hoh BG, Hunte HER, Marshall M, Mohile SG, Plumb S, Tejani MA, Venuti A, Epstein RM. The social and behavioral influences (SBI) study: study design and rationale for studying the effects of race and activation on cancer pain management. BMC Cancer. 2017 Aug 25;17(1):575. doi: 10.1186/s12885-017-3564-2. PMID 28841847